CLINICAL TRIAL: NCT02771496
Title: ROCK Comprehensive Prospective Cohort for Osteochondritis Dissecans of the Knee
Brief Title: Osteochondritis Dissecans of Knee Prospective Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Altona Children's Hospital (Other); Boston Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Health Andrews Institute for Orthopaedics & Sports Medicine (Unknown); Children's Healthcare of Atlanta (Other); Children's Hospital Colorado (Other); Children's Hospital of Philadelphia (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Children's Mercy Hospital Kansas City (Other); Connecticut Children's Medical Center (Other); Hospital for Special Surgery, New York (Other); Kaiser Permanente (Other); Mayo Clinic (Other); National University Hospital, Singapore (Other); Rady Children's Hospital, San Diego (Other); Stanford University (Other); Tennessee Orthopedic Alliance (Other); Texas Scottish Rite Hospital for Children (Other); The Rocky Mountain Hospital for Children (Unknown); The Hospital for Sick Children (Other); Göteborg University (Other); University of Minnesota/TRIA Orthopaedic Center (Unknown); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 820147
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Osteochondritis Dissecans
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with OCD: Patients with diagnosis of OCD as confirmed by x-ray or MRI. Surveys collected from patients at 2 years, 5 years, 10 years, and 25 years.
  Interventions: Other: Other: observational only- no intervention

INTERVENTIONS:
Other: Other: observational only- no intervention — Other: observational only- no intervention

SUMMARY:
The Cohort is a multi-site prospective data collection study that will enroll any patient with diagnosis of knee OCD (confirmed by a standard of care x-ray or MRI). Patients will be followed for up to the next 50 years of their lives to study courses of care, disease progression, treatment/surgical options/results, and specific sports-related outcomes in athletic patients. Subjects will complete quality of life surveys as part of the Cohort. Course of care will not be affected.

DETAILED DESCRIPTION:
Patients will be recruited and consented at the visit in which their eligibility is determined. Once a patient is eligible and provides informed consent, he or she will be in the study for up to 50 years, or until his or her OCD lesion is healed successfully.

At the initial visit, a subject will complete a basic medical history form, and three questionnaires: the IKDC Subjective questionnaire (ages over 18) or the PEDI-IKDC Subjective questionnaire (ages under 18); the KOOS questionnaire; and the Marx Activity Scale (adult) or Pedi-FABS Scale (pediatric). Patients will then continue with their normal course of care as determined by their surgeon and care team.

Mandatory surveys (same as above) will be collected from patients at 2 years, 5 years, 10 years, and 25 years. Patients who cannot return to clinic will have the option to complete the assessments and return in pre-stamped and addressed return envelopes provided by the clinical site the subject is a patient at. Any other follow-up visits between these time intervals will also be options for patients to complete these assessments, however patients will not complete them any closer than intervals 12 weeks apart in order to prevent redundancy.

Additionally, at the initial visit, the surgeon will complete a routine patient history and physical exam, which will be collected. Any surgical procedures or physical therapy a patient undergoes for treatment of his or her OCD lesion will also be documented and collected. At follow-up visits, surgeons will complete their own physical exam follow-up assessment forms, which will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteochondritis dissecans or focal articular cartilage defects as confirmed by x-ray or MRI

Exclusion Criteria:

* Non-confirmed diagnosis (i.e. patient does not yet have imaging confirmation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages with osteochondritis dissecans (OCD) or focal articular cartilage defects confirmed via MRI or x-ray.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2014-05; Primary Completion 2064-05 (Estimated); Study Completion 2064-12 (Estimated)

PRIMARY OUTCOMES:
IKDC questionnaire | baseline up to 50 years
  The primary outcome endpoint for this study is the patient's score on the IKDC Subjective questionnaire, or PEDI-IKDC Subjective questionnaire for patients under 18 years of age.
PEDI-IKDC questionnaire | baseline up to 50 years
  The primary outcome endpoint for this study is the patient's score on the IKDC Subjective questionnaire, or PEDI-IKDC Subjective questionnaire for patients under 18 years of age.

SECONDARY OUTCOMES:
KOOS Knee score | baseline up to 50 years
  The Knee injury and Osteoarthritis Outcome Score (KOOS) evaluates short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis.
Marx Activity Score questionnaire | baseline up to 50 years
  Measure of physical activity at healthiest and most active state from time of taking to year prior.
Pedi-FABS Score | baseline up to 50 years
  An eight-item scale that measures level of physical activity and fitness.
Radiographic Healing | baseline up to 50 years
  Visualization of bone healing through x-ray images.

CONTACTS AND LOCATIONS:
Overall Officials: James L Carey, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided